CLINICAL TRIAL: NCT04642313
Title: Comparison of Magnesium Versus Potassium and Their Combined Effect on Insomnia, Sleep Hormones, Insulin Resistance and Quality of Life Among Patients With Diabetes Mellitus".
Brief Title: Comparison of Mg Vs. K Supplementation on Insomnia in Diabetics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Sidra Khalid, PhD Scholar, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL-UIDNS-Mg-K
Record Dates: First submitted 2020-11-09; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Focus of Study is on Insomnia Among Diabetic Patients
Keywords: Insomnia, Diabetes Mellitus, Magnesium, Potassium, Melatonin, Cortisol, Insulin resistance, Quality of Life
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Diabetes Mellitus; Insulin Resistance | interventions — Magnesium; Potassium

STUDY DESIGN:
Intervention Model Description: Participants will be divided into 4 groups and will receive 4 different treatments at same time
Who Masked: Participant
Masking Description: It will be single blind study, Participants will not be aware of the treatment group, they are receiving
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PLACEBO group (Placebo Comparator): Placebo treatment: starch tablets (250 mg)
  Interventions: Other: Magnesium and/ or Potassium
- Magnesium group (Experimental): Magnesium group: Magnesium gluconate (250 mg)
  Interventions: Other: Magnesium and/ or Potassium
- Potassium group (Experimental): Potassium group: Potassium chloride (250 mg)
  Interventions: Other: Magnesium and/ or Potassium
- Magnesium + Potassium group (Experimental): Magnesium + Potassium group: Magnesium gluconate (250 mg) + Potassium chloride (250 mg)
  Interventions: Other: Magnesium and/ or Potassium

INTERVENTIONS:
Other: Magnesium and/ or Potassium — Magnesium and/ or potassium supplements will be provided to patients of diabetes mellitus with insomnia

SUMMARY:
Insomnia is increasing alarmingly among the population. Micronutrient fluctuations have been shown to effect insulin secretion, period of circadian cycle and quality of sleep in all ages. This study is aimed to identify the impact of magnesium and potassium supplementation on insomnia severity and duration, and insulin resistance, quality of life, sleep hormones, serum magnesium and potassium levels. Moreover, the study will help to find out the link between insomnia and micronutrients among patients of diabetes mellitus so that the burden of the disease in the society could be reduced.

DETAILED DESCRIPTION:
Sleep is the essential component to maintain good health of an individual. Insomnia is defined as a condition that affects an individual by inability to get sufficient quality sleep or problem in maintaining sleep that is important for healthy functioning, performance and well being. Insomnia can exist in healthy individual or comorbidly with other medical diseases. Latest researches indicate that intolerance of glucose in the body, resistance to insulin hormone, decreased acute response of insulin to glucose and increased chances of having type 2 diabetes are reasons for reduced or interrupted sleep. Several electrolytes and minerals influence the sleep cycle. Magnesium is important in regulation of central nervous system excitability, through ion channel conductivity. Magnesium is a muscle relaxant and inducer of the deeper sleep. Hypomagnesemia is a common feature in patients with type 2 diabetes. Although diabetes can induce hypomagnesemia, magnesium deficiency has also been proposed as a risk factor for type 2 diabetes. Magnesium supplementation improves sleep efficiency, sleep time and sleep onset latency, early morning awakening, and insomnia objective measures such as the concentration of serum renin, melatonin, and serum cortisol, in older adults. High ambient potassium levels have been shown to shorten the period of circadian rhythms in a variety of organisms. Little is known about the effects of dietary mineral nutrients on human sleep quality. Potassium depletion has been shown to cause glucose intolerance, which is associated with impaired insulin secretion . Recently, there has been growing evidence from both animal and human studies indicating that high sodium and low potassium intakes are associated with a high risk of insulin resistance or diabetes.

The Study is aimed to:

1. To compare the effect of magnesium and/ or potassium on insomnia patients with diabetes mellitus
2. To compare the gender and age based response to magnesium and/ or potassium on insomnia patients with diabetes mellitus
3. To compare the effect of magnesium and/ or potassium on insulin resistance among insomnia patients with diabetes mellitus
4. To compare the effect of magnesium and/ or potassium on sleep hormones among insomnia patients with diabetes mellitus
5. To compare the effect of magnesium and/ or potassium on serum electrolytes (Mg, K) among insomnia patients with diabetes mellitus
6. To compare the effect of magnesium and/ or potassium on quality of life (QOL) among insomnia patients with diabetes mellitus MATERIAL AND METHODS Study Design: Randomized Controlled Trial (single blind) Settings: Study will be conducted at

1. Akhuwat Health Services, Lahore Duration of Study: 18 months (after the approval of synopsis) Sample Size: is 280 and with expected 20% drop out: 320 Sampling Technique: Non probability purposive sampling

Inclusion Criteria:

* Patients of diabetes mellitus with insomnia
* Adult diabetic patients aged between 19 to 65 years
* Patients of both genders
* Diabetic patients of insomnia with or without antidiabetic drugs

ELIGIBILITY:
Inclusion Criteria:

* • Patients of diabetes mellitus with insomnia

  * Adult diabetic patients aged between 19 to 65 years
  * Patients of both genders
  * Diabetic patients of insomnia with or without anti-diabetic drugs
  * Diabetic patients of insomnia with or without Hypomagnesaemia
  * Diabetic patients of insomnia with or without Hypokalemia

Exclusion Criteria:

* Individuals with the following conditions will not be included as participants, patients of diabetes mellitus with insomnia with

  * Psychiatry reasons
  * Any hormonal treatment
  * CVD/ Other metabolic co-morbidities
  * History of acute liver injury (e.g., hepatitis) or severe cirrhosis
  * Renal diseases (renal stones, renal failure, dialysis)
  * Diabetic nephropathy
  * Pregnancy
  * Breast-feeding
  * Drug induced insomnia
  * Sleep disorders
  * Sleep-related movement disorders (restless leg syndrome)
  * Sleep-related respiratory disorders (sleep apnea)
  * Alcohol consumption
  * Cardiac respiratory disorders
  * Painful condition (apathy)
  * History of chronic liver disease
  * History of CKD
  * Participation in a study of an investigational medication or nutritional supplements/ medication within the past 90 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-04-26 (Estimated); Study Completion 2022-04-26 (Estimated)

PRIMARY OUTCOMES:
Effects of magnesium and/ or potassium supplementation on insomnia severity patients with diabetes mellitus | 60 days
  Insomnia Severity Index (ISI) will be used to assess and categorize the insomnia among patients with diabetes mellitus, before and after the intervention
Effects of magnesium and/ or potassium on insulin resistance among insomnia patients with diabetes mellitus | 60 days
  Homeostatic model assessment for insulin resistance (HOMA-IR) will be used to measure the insulin resistance before and after the Mg, K supplementation among insomniac patients with diabetes mellitus. Insulin will be measured through ELISA technique.
Effects of magnesium and/ or potassium on sleep hormones (melatonin, cortisol) among insomniac patients with diabetes mellitus. | 60 days
  Sleep hormones (melatonin, cortisol) will be measured before and after the intervention, through ELISA technique, among insomniac patients with diabetes mellitus.
Effect of magnesium and/ or potassium on serum electrolytes (Mg, K) among insomnia patients with diabetes mellitus | 60 days
  Serum magnesium and/ potassium (in blood) will be measured through chemistry analyzer, before and after the Mg, K supplementation among insomniac patients with diabetes mellitus

SECONDARY OUTCOMES:
Effect of magnesium and/ or potassium on quality of life (QOL) among insomnia patients with diabetes mellitus | 60 days
  WHOQOL-BREF will be used to measure quality of life before and after the Mg, K supplementation, among insomniac patients with diabetes mellitus.
Gender and age based response to magnesium and/ or potassium on insomnia patients with diabetes mellitus | 60 days
  Gender and age based responses of Mg, K supplementation will be compared among insomniac patients with diabetes mellitus

OTHER OUTCOMES:
Effect of magnesium and/ or potassium on quality liver function tests (LFTs) among insomnia patients with diabetes mellitus | 60 Days
  Liver function tests (ALT, AST) will measured before and after the Mg, K supplementation among insomniac patients with diabetes mellitus

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Akhuwat Health Services, Lahore, Punjab Province
  - The University of Lahore, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No
Patients data will be kept confidential and their identity will not be revealed

REFERENCES:
- [Derived] Khalid S, Mehboob R, Bokhari SS, Ali M, Shabbir A, Mehboob K, Adnan H, Karami MM, Shalabi H, Alshehri B. Comparative Efficacy of Magnesium and Potassium Towards Cholesterol and Quality of Life in Patients With Type 2 Diabetes Mellitus: A Randomised Single-Blinded Controlled Clinical Trial. Endocrinol Diabetes Metab. 2024 Nov;7(6):e511. doi: 10.1002/edm2.511. PMID 39410716